CLINICAL TRIAL: NCT00297843
Title: A Pilot Monocenter Study to Assess the Reproducibility and Specificity of Cellular and Soluble Biomarkers in Nasal Secretions in Patients With Allergic Rhinitis and Healthy Volunteers Following Pollen Exposure in the Fraunhofer Environmental Challenge Chamber (ECC)
Brief Title: A Pilot Monocenter Study to Assess Cellular and Soluble Biomarkers in Nasal Secretions
Status: Completed | Type: Observational
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Other Study IDs: 06/01 Nabio ITEM
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-06

CONDITIONS: Seasonal Allergic Rhinitis; Healthy Subjects
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Nasal Lavage

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Procedure: allergen challenge (grass pollen), nasal lavage

SUMMARY:
Allergic Rhinitis is an inflammatory disease which causes an influx of inflammatory cells and cytokines into the nasal mucosa. These biomarkers can also be found in the nasal secretions. The evaluation of these inflammatory biomarkers is of great interest as this could lead to a concept of measuring the efficacy of anti-allergic treatments by assessing the changes in nasal biomarkers after allergen challenge. To use this model as an assessment of pharmacodynamics it is crucial to evaluate the specificity and reproducibility of cellular and cytokine levels in the nasal secretions after allergen provocations.

In a 2 part repeated measurement design 20 patients with allergic rhinitis and 20 healthy subjects will undergo two 4-hour pollen exposures in an interval of 21 days.

The aim of this study is to explore the cellular and cytokine levels this allergen challenge will induce in nasal secretions and to assess if an increase in those inflammatory biomarkers is specific to the patient subgroup and whether the results are reproducible after the second allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-55 years.
* Women will be considered for inclusion if they are: Not pregnant or nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and have been amenorrhoeic for more than 1 year prior to the screening visit).Of childbearing potential and using an appropriate method of contraception (Oral contraceptive pill or double barrier).
* FEV1 > 80% of predicted at screening.
* Absence of any structural nasal abnormalities or nasal polyps on examination, a history of frequent nose bleeding or recent nasal surgery.
* Absence of conditions or factors, which would make the subject unlikely to be able to stay in the Fraunhofer ECC for 4 hours.
* Non smoker or smokers with a history of less than 10 pack years.
* Able and willing to give written informed consent to take part in the study.
* Available to complete all study measurements.
* For subjects with allergic rhinitis:
* History of allergic rhinitis to grass pollen and a positive skin prick test for Dactylis glomerata pollen at or within 12 months prior to the screening visit.
* Subject must exhibit a moderate response upon 4.000 Dactylis glomerata pollen grains/m3 during 4 hours in the ECC on visit 2, which is defined as a Total Nasal Symptom Score of at least 6. (TNSS is the sum of obstruction, rhinorrhea, itch, and sneeze, each of which has been scored on a scale from 0 to 3).
* Subjects with mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function may be included also.
* Total Nasal Symptom Score (TNSS) of < 3 and a score < 2 for each symptom, i.e. obstruction, rhinorrhea, itch, and sneeze prior to entering the pollen chamber.
* for healthy subjects:
* No history of allergic rhinitis and a negative skin prick test including Dactylis glomerata at or within 12 months prior to the screening visit.
* Total Nasal Symptom Score (TNSS) prior to and during pollen exposition of < 3 and a score < 2 for each symptom, i.e. obstruction, rhinorrhea, itch, and sneeze.
* Absence of any respiratory disease

Exclusion Criteria:

* History of a respiratory tract infection and/or exacerbation of asthma within 4 weeks before the informed consent and during the study.
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest or hypoxic seizures.
* Administration of oral, injectable or dermal corticosteroids within 8 weeks or intranasal and/or inhaled corticosteroids within 4 weeks of the screening visit.
* Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDS), anti-depressant drugs, anti-histamines and anti-asthma, anti-rhinitis or hay fever medication (other than short acting inhaled beta-agonists) and paracetamol (up to 1g paracetamol per day is permitted for the treatment of minor ailments e.g. headache) for 1 week prior to screening and throughout the course of the study.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Subject is undergoing allergen desensitisation therapy
* There is a risk of non-compliance with study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-03; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, MD, Principal Investigator — Fraunhofer ITEM, Nikolai-Fuchs-Str. 1, 30625 Hannover, Germany
Locations (1):
- Fraunhofer ITEM, Hanover, Germany

REFERENCES:
- [Derived] Badorrek P, Muller M, Koch W, Hohlfeld JM, Krug N. Specificity and reproducibility of nasal biomarkers in patients with allergic rhinitis after allergen challenge chamber exposure. Ann Allergy Asthma Immunol. 2017 Mar;118(3):290-297. doi: 10.1016/j.anai.2017.01.018. PMID 28284536